CLINICAL TRIAL: NCT05440539
Title: Educating Women About Pelvic Floor Disorders During Pregnancy From the 1st to the "4th Trimester": A Randomized Clinical Trial
Brief Title: Educating Women About Pelvic Floor Disorders During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PFD Education in Pregnancy
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Floor Disorders; Stress Urinary Incontinence; Pelvic Organ Prolapse
Keywords: pregnancy; education; prolapse; incontinence
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence, Stress; Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Group (Experimental): Participants received only written handouts with information about pelvic floor disorders, including risk factors, prevention strategies, and information about possible treatments. They receive these handouts at the time of recruitment during pregnancy and again after delivery.
  Interventions: Other: Written Handouts
- Workshop Group (Experimental): Participants received written handouts and attend a virtual interactive workshop with information about pelvic floor disorders, including risk factors, prevention strategies, and information about possible treatments. They receive the handouts at the time of recruitment during pregnancy and again after delivery. The workshop is conducted prior to completion of pregnancy.
  Interventions: Other: Written Handouts; Other: Interactive Workshop

INTERVENTIONS:
Other: Written Handouts — The written materials were generated using the collaboration of healthcare communication specialists to generate content that is tailored to a younger age demographic of childbearing age regarding their risk of developing a pelvic floor disorder and what can be done to prevent or treat them in the future.
Other: Interactive Workshop — Participants logged onto a virtual meeting platform and listened to a live 20 minute presentation by a pelvic floor physical therapist followed by time for questions, which were answered live. Participants anonymity was maintained by not allowing participants to view each other's name and disabling sharing of video feeds.
  Arms: Workshop Group

SUMMARY:
The purpose of this study is to assess the increase in knowledge of pregnant patients regarding pelvic floor disorders when comparing two educational interventions: written handouts vs interactive workshops.

DETAILED DESCRIPTION:
Pelvic floor disorders (PFDs) are common and significantly affect the quality of life of many women as they age. Pregnancy has been identified as a major risk factor for developing PFDs later in life. Educating women about PFDs is essential to ensuring that they present to care in a timely manner. No study has investigated different education tools during pregnancy. The proposed study is a randomized controlled trial in pregnant patients comparing two educational tools: written materials about PFDs versus an educational workshops led by pelvic floor physical therapists (PFPTs). Pregnant patients will be recruited in the first and second trimester and randomized at that time. Knowledge will be assessed at baseline and again 6 weeks postpartum using the validated Prolapse and Incontinence Knowledge Questionnaire. Secondary outcomes will be evaluating referral patterns to urogynecology and to PFPTs from general OBGYNs and assessing any pelvic floor symptoms with the pelvic floor disability index (PFDI-20) at baseline and at 6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (prior to 27 weeks gestation)
* English speaking
* Greater than 18 years old

Exclusion Criteria:

* Non-english speaking
* unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durnea CM, Khashan AS, Kenny LC, Durnea UA, Dornan JC, O'Sullivan SM, O'Reilly BA. What is to blame for postnatal pelvic floor dysfunction in primiparous women-Pre-pregnancy or intrapartum risk factors? Eur J Obstet Gynecol Reprod Biol. 2017 Jul;214:36-43. doi: 10.1016/j.ejogrb.2017.04.036. Epub 2017 Apr 23. PMID 28525825
- [Background] McLennan MT, Melick CF, Alten B, Young J, Hoehn MR. Patients' knowledge of potential pelvic floor changes associated with pregnancy and delivery. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Jan;17(1):22-6. doi: 10.1007/s00192-005-1325-2. Epub 2005 Jul 8. PMID 16003482
- [Background] Koury H, Corral J, Bastow BD, Sheeder J, Muffly TM. A 3-Dimensional Anatomical Education Model in Postpartum Perineal Laceration Care: A Pre-Post Intervention Study. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):e23-e27. doi: 10.1097/SPV.0000000000000698. PMID 30807431
- [Background] Gagnon LH, Boucher J, Robert M. Impact of pelvic floor muscle training in the postpartum period. Int Urogynecol J. 2016 Feb;27(2):255-60. doi: 10.1007/s00192-015-2822-6. Epub 2015 Aug 19. PMID 26282094
- [Background] Shah AD, Massagli MP, Kohli N, Rajan SS, Braaten KP, Hoyte L. A reliable, valid instrument to assess patient knowledge about urinary incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Sep;19(9):1283-9. doi: 10.1007/s00192-008-0631-x. Epub 2008 May 15. PMID 18480958
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Haller J, Keller Z, Barr S, Hadden K, Oliphant SS. Assessing Readability: Are Urogynecologic Patient Education Materials at an Appropriate Reading Level? Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):139-144. doi: 10.1097/SPV.0000000000000653. PMID 30807416
- [Derived] Rutledge E, Spiers A, Vardeman J, Griffin N, Nisar T, Muir T, Antosh DD. Educating Women About Pelvic Floor Disorders During Pregnancy From the First to the "Fourth Trimester": A Randomized Clinical Trial. Urogynecology (Phila). 2023 Sep 1;29(9):770-776. doi: 10.1097/SPV.0000000000001341. PMID 37607311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited between August 2020 and Sept 2021. Patients were identified via medical records and approached in an obstetrics clinic at a single institution.
Pre-assignment Details: Participants were excluded if they were not english speaking or were unable to give consent due to being a minor or unable to provide consent.
Period: Overall Study
Arm/Group | Written Group | Workshop Group
Started | 61 | 59
Completed | 54 | 51
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 4 | 4
Not completed — Fetal demise, no longer pregnant | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Written Group | Workshop Group | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 32 [30 to 37] | 32 [29.5 to 35] | 32 [19 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 120
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 32 | 60
  Hispanic | 20 | 13 | 33
  Black | 8 | 7 | 15
  Asian | 4 | 7 | 11
  Other (unspecified) | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 120
Income Level [Count of Participants; unit: Participants]
  <10,000 | 1 | 5 | 6
  10,000-49,999 | 6 | 5 | 11
  50,000-100,000 | 16 | 13 | 29
  >100,000 | 38 | 36 | 74
Gravida [Median (Inter-Quartile Range); unit: Number of Pregnancies] | 1 [1 to 2.5] | 2 [1 to 3] | 2 [1 to 6]
Para [Median (Inter-Quartile Range); unit: Number of Deliveries] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 5]
Pre-Pregnancy BMI [Median (Inter-Quartile Range); unit: kg/m2] | 27.1 [24.1 to 30.9] | 25.5 [22.65 to 30.35] | 26.2 [19.6 to 55.8]
Married [Count of Participants; unit: Participants] | 47 | 50 | 97
Education Level [Count of Participants; unit: Participants]
  High School | 3 | 7 | 10
  College | 32 | 25 | 57
  Graduate School | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Prolapse and Incontinence Knowledge Questionnaire (PIKQ)
Description: Validated 24 question questionnaire with two sections to test knowledge on pelvic organ prolapse and urinary incontinence. Scored out of 24 with higher scores indicating an increase in knowledge. Minimum value: 0, Maximum value: 24. Higher scores mean better outcome. Lower scores mean worse outcome. This was administrated at time of recruitment and again at 6 weeks postpartum.
Time Frame: < 5 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Written Group | Workshop Group
Number analyzed (Participants) | 61 | 59
score on a scale
  Pre-PIKQ | 17 [14 to 22] | 17 [13 to 20]
  Post-PIKQ | 21 [19 to 23] | 21 [17 to 22]

2. Secondary Outcome: Pelvic Floor Distress Inventory (PFDI-20)
Description: Validated questionnaire measuring presence and degree of both of pelvic floor disorder symptoms. Three sub sections with a possible score of 100 for each sub section. Scaled score is a combination of the 3 sub section scores for a total possible score of 300. Higher scores indicates increased symptom bother. Minimum value: 0, Maximum value: 300. Higher scores mean better outcome. Lower scores mean worse outcome. This was administrated at time of recruitment and again at 6 weeks postpartum.
Time Frame: < 5 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Written Group | Workshop Group
Number analyzed (Participants) | 61 | 59
score on a scale
  Pre-PFDI | 29.17 [12.50 to 64.58] | 36.47 [17.71 to 62.50]
  Post-PFDI | 14.58 [0 to 25] | 9.89 [3.13 to 22.92]

3. Secondary Outcome: Phone Interview
Description: One-on-one phone interviews conducted with participants in the workshop education group who experienced both educational tools. A research team member called them after completion of the study and conducted a brief 3 question interview to understand their opinion of the educational tools.
Time Frame: < 10 minutes
Population: Only the workshop group were included in the phone interview portion of the study as they experienced both interventions: written handouts and virtual workshop.
Measure: Count of Participants; unit: Participants
Arm/Group | Written Group | Workshop Group
Number analyzed (Participants) | 0 | 34
Participants
  Preferred workshop format |  | 20
  Preferred written format |  | 14

ADVERSE EVENTS:
Time Frame: August 2020 until September 2021 Participants were recruited in the 1st and 2nd trimester of pregnancy and remained in the study until 6 weeks postpartum. The estimated time of involvement in the study was between 6-8 months depending on the point in pregnancy at which they were recruited.
Arm/Group | Written Group | Workshop Group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 0/61 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05440539/Prot_SAP_000.pdf